CLINICAL TRIAL: NCT04824456
Title: Evaluation of Neurosensory Disturbance After Using Separators Vs Chisels in Bilateral Sagittal Split Mandibular Osteotomy. RCT
Brief Title: Neurosensory Assesment After Using Separators Vs Chisels in Bilateral Sagittal Split Mandibular Osteotomy. RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hisham Mohammed Abdllfattah, Assistant lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 15460
Record Dates: First submitted 2020-11-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: to Assess Neurosensory Function of Inferior Alveolar Nerve After BSSO

STUDY DESIGN:
Intervention Model Description: Patient with skeletal malocclusion, class II or class III that is indicated for bilateral sagittal split osteotomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bilateral sagittal split osteotomy using chisels. (Experimental): The final split is completed with Smith forceps and flag separators
  Interventions: Procedure: bilateral sagittal split osteotomy using separators.

INTERVENTIONS:
Procedure: bilateral sagittal split osteotomy using separators. — The final split is completed with a thin osteotomes, splitting the entire ascending ramus from the anterior to the posterior border of the ramus.

SUMMARY:
The bilateral sagittal split Ramus osteotomy (BSSRO) was introduced by Trauner and Obwegeser. Since then, many modifications of this procedure have been reported, leading to a less difficult and more predictable procedure for correcting mandibular anomalies. persistent post-operative neurosensory disturbances of the inferior alveolar nerve are still one of the major complications of this operation. The incidence has decreased over the years due to improved techniques and the use of different instruments. However, most recent series still report postoperative persistent hypesthesia of the inferior alveolar nerve in more than 10% of the patients up to 48%.

There are no reports on the influence of other surgical variables on the persisting post-operative hypesthesia. Several methods have been reported for evaluating neurosensory disturbances of the inferior alveolar nerve. One of the simplest methods reported is tactile evaluation based on subjective sensation reported by the patients. Many authors have used this method in their evaluation of post-operative hypesthesia.

ELIGIBILITY:
IInclusion criteria:

1. Patient with skeletal malocclusion, class II or class III that is indicated for bilateral sagittal split osteotomy.
2. Adults >18 years.
3. Systemically healthy.

Exclusion criteria:

1. Patients not indicated for orthognathic surgery.
2. Severe systemic disease.
3. Have a medical condition associated with systemic neuropathy (e.g. diabetes)
4. Patients whom cannot tolerate follow up intervals. (affect accuracy of study results)
5. Are unwilling to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
neurosensory disturbance of the inferior alveolar nerve. | 1 year
  use Von Frey filaments to test sensory function of the lower lip and two point discrimination test (blunt and sharp ) also to assess the sensory function

SECONDARY OUTCOMES:
Incidence of bad split | 1 year
  if bad split in the mandible occur during the operation it will be reported
post operative edema , | 1 year
  preoperative measure from the tragus to mid of the chin by cm then the measure is repeated to count the amount of edema
post operative pain | 1 year
  by visual analogue scale from 0 to 10 and the patient choose the number

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No